CLINICAL TRIAL: NCT07067736
Title: Cefazolin Antibiotic Prophylaxis in Ventricular Shunt Surgery: Determination of Cerebrospinal Fluid(CSF) Concentration During Valve Implantation
Brief Title: Cefazolin Antibiotic Prophylaxis in Ventricular Shunt Surgery: Determination of Cerebrospinal Fluid Concentration During Valve Implantation
Acronym: CC -PIV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 9720
Record Dates: First submitted 2025-06-24; First posted 2025-07-16 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Hydrocephaly; CSF Shunts; Antibiotic Prophylaxis
Keywords: Antibiotic prophylaxis; CSF shunts; Hydrocephaly
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cefazolin antibiotic prophylaxis in ventricular shunt surgery (Experimental)
  Interventions: Other: Cefazolin antibiotic prophylaxis

INTERVENTIONS:
Other: Cefazolin antibiotic prophylaxis — Determination of cerebrospinal fluid concentration

SUMMARY:
The objective is to determine the concentration of cefazolin in the cerebrospinal fluid after a recommended antiobiotic prophylaxis by 2g of cefazolin. Our main hypothesis is that the concentration is insufficient to protect the valve from infections.

The secondary objective is to compare our results to known pharmacokinetic models of cefazolin diffusion in the literature. If differences are found we would like to search clinical features that could explain it.

ELIGIBILITY:
Inclusion Criteria:

Age >18 years and programmed for a ventricular shunt surgery at the Hautepierre university hospital in Strasbourg.

Exclusion Criteria:

* Age <18 years old
* Pregnant women
* Infected patients
* Known cefazolin allergy
* Other molecule used for the antibiotic prophylaxis
* Guardianship or conservatorship
* Patients under curative antibiotherapy
* Non sterile pre operative CSF
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Cefazolin concentration in the cerebrospinal fluid | The measure is made when the dura mater is opened just before the valve implantation.
  Cefazolin concentration in the cerebrospinal fluid.

SECONDARY OUTCOMES:
blood cefazolin concentration | Blood samples are made before injection
  Compare the cerebrospinal and blood cefazolin concentration to the known pharmacokinetic models in order to determine clinical features that could explain thoses differences.
blood cefazolin concentration | Blood samples are made 30 minutes , after injection
  Compare the cerebrospinal and blood cefazolin concentration to the known pharmacokinetic models in order to determine clinical features that could explain thoses differences.
blood cefazolin concentration | Blood samples are made 1hour after injection
  Compare the cerebrospinal and blood cefazolin concentration to the known pharmacokinetic models in order to determine clinical features that could explain thoses differences.
blood cefazolin concentration | Blood samples are made 2 hours after injection
  Compare the cerebrospinal and blood cefazolin concentration to the known pharmacokinetic models in order to determine clinical features that could explain thoses differences.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No